CLINICAL TRIAL: NCT03790709
Title: A Phase 2b/3, Double-Blind, Randomized, Placebo-Controlled 48-week Safety and Efficacy Trial of ANAVEX2-73 for the Treatment of Early Alzheimer's Disease (AD)
Brief Title: ANAVEX2-73 for Treatment of Early Alzheimer's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Anavex Life Sciences Corp. (Industry)
Collaborators: Anavex Australia Pty Ltd. (Industry); Anavex Germany GmbH (Industry); Anavex Canada Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAVEX2-73-AD-004
Record Dates: First submitted 2018-12-24; First posted 2019-01-02 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tetrahydro-N, N-dimethyl-2,2-diphenyl-3-furanmethanamine hydrochloride

STUDY DESIGN:
Intervention Model Description: Randomized 1:1:1 to two different ANAVEX2-73 doses or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There will be blinding procedures for this study. Capsules will be indistinguishable from active ingridient containing capsules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose ANAVEX2-73 (Experimental): High dose active once daily orally
  Interventions: Drug: High dose ANAVEX2-73
- Mid dose ANAVEX2-73 (Experimental): Mid dose active once daily orally
  Interventions: Drug: Mid dose ANAVEX2-73
- Placebo oral capsule (Placebo Comparator): Placebo dose once daily orally
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: High dose ANAVEX2-73 — Oral capsule
  Arms: High dose ANAVEX2-73
Drug: Mid dose ANAVEX2-73 — Oral capsule
  Arms: Mid dose ANAVEX2-73
Drug: Placebo oral capsule — Oral capsule
  Arms: Placebo oral capsule

SUMMARY:
Phase 2b/3 48-week study to evaluate the effects of ANAVEX2-73 on cognition and function after 48 weeks of daily treatment. Additional outcome measures include refined measures of sleep, behavioral and psychological symptoms typically observed in AD, changes in daily functioning of participants and changes in caregiver burden, as well as changes in quality of life measures of both, patients and caregivers during treatment with ANAVEX2-73.

DETAILED DESCRIPTION:
This is a Phase 2b/3 48-week study to evaluate the effects of ANAVEX2-73 on cognition and function after 48 weeks of daily treatment. Additional outcome measures include refined measures of sleep, behavioral and psychological symptoms typically observed in AD, changes in daily functioning of participants and changes in caregiver burden, as well as changes in quality of life measures of both, patients and caregivers during treatment with ANAVEX2-73. In addition, safety assessments, pharmacokinetic (PK) assessments and collections of CSF and blood markers of AD pathophysiology before and after treatment will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 to 85 years, inclusive, with a NIA-AA diagnosis of mild cognitive impairment (MCI) due to AD or early stage mild dementia due to AD. AD diagnosis should be made by an appropriately qualified medical specialist and AD pathology should be confirmed by either:

  1. Historical records of amyloid CSF assessment or
  2. Historical records of amyloid PET scan or
  3. If neither historical records are available, then AD pathological diagnosis confirmation should be offered at screening:

  i. CSF collection or ii. Amyloid PET iii. Past medical records of MRI or CT are optional.
* Mini Mental State Examination (MMSE) score between 20-28, inclusive.
* Free Recall score ≤17 or Total Recall score <40 on the Free and Cued Selective Reminding Test (FCSRT).
* Participants are either outpatients, or residents of an assisted-living facility. Participant has a designated study partner, who spends at least 10hrs per week with the participant, in order that assessments e.g. carer burden instruments are completed with true knowledge of the participant.
* No suicidal ideation of type 4 or 5 in the Columbia Suicide Severity Rating Scale (C-SSRS) in the past 3 months (i.e. active suicidal thought(s) with intent but without specific plan, or active suicidal thought(s) with plan and intent) OR suicidal behavior in the past 2 years (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior).
* Confirmation from the participant that, if of childbearing potential is not pregnant through urine pregnancy testing.

Exclusion Criteria:

* Patients who have a progressive medical or neurological condition that in the opinion of the investigator would interfere with the conduct of the study. Exception: If diagnosed with seizures, must be on stable anti-seizure medication for at least 3 months prior to screening.
* Current clinically significant systemic illness that is likely to result in deterioration of the patient's condition or affect the patient's safety during the study.
* History or clinically evident stroke or clinically significant carotid or vertebrobasilar stenosis or plaque.
* History of neurologic (e.g. stroke, traumatic brain injury) or psychiatric condition that the investigator deems may interfere with interpretability of data.
* History of untreated thyroid disorder, Type 1 diabetes, and insulin dependent or uncontrolled Type II diabetes, as determined by the investigator (e.g. non-insulin-controlled Type II diabetes, whose HbA1c value is higher than 8.0%).
* Body Mass Index (BMI) > 30.
* History of clinical hepatic dysfunction.
* Current symptomatic and unstable/uncontrolled gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, hematological or hormonal disorders.
* Indication of liver disease, defined by serum levels of ALT (SGPT), AST (SGOT), or alkaline phosphatase above 3x upper limit of normal (ULN) as determined during screening.
* Significant history of drug addiction (with the exception of nicotine dependence) or abuse (including alcohol, as defined in DSM-V or in the opinion of the investigator) within the last two years prior to informed consent, or a positive urine drug screen for cocaine, opioid, phencyclidine (PCP), amphetamine or marijuana at screening. Prescription medication yielding a positive drug screen are acceptable except for tricyclic antidepressants (e.g. Amitriptyline, Amoxapine, Desipramine, (Norpramin) Doxepin, Imipramine (Tofranil), Nortriptyline (Pamelor), Protriptyline (Vivactil), Trimipramine (Surmontil)).
* Clinically significant infection within the last 30 days prior screening (e.g., chronic persistent or acute infection, urinary tract infections (UTI)).
* Treatment with immunosuppressive medications (e.g., systemic corticosteroids) within the last 90 days (topical and nasal corticosteroids and inhaled corticosteroids for asthma are permitted) or chemotherapeutic agents for malignancy within the last 3 years.
* Myocardial infarction within the last year.
* History of cancer within the last 3 years, with the exception of basal cell carcinoma and non-metastatic squamous cell carcinoma of the skin and prostate cancer with currently normal PSA.
* Other clinically significant abnormality on physical, neurological, laboratory, or electrocardiogram (ECG) examination (e.g., atrial fibrillation) that could compromise the study or be detrimental to the participant.
* Hemoglobin < 11 g/dL.
* Have any contraindication to MRI scanning, including cardiac pacemaker/defibrillator, ferromagnetic metal implants (e.g., in skull and cardiac devices or severe claustrophobia).
* Smoking > 1 pack of cigarettes per day (as assessed for the 30 days prior to screening).
* Alcohol use of more than 2 drinks per day.
* Current use of over-the-counter (OTC) supplements or nutraceuticals unless they are on stable dose for at least 3 months prior to screening and are documented in the eCRF.
* Use of over the counter (OTC) or prescription medication for sleep on 2 or more occasions per week.
* Being treated with psychoactive medications on a stable dose for less than 3 month.
* Any prior exposure to ANAVEX2-73.
* Individuals enrolled in previous AD clinical trial involving an investigational drug treatment less than 3 months ago (longer than 3 month ago allowed).
* Any known hypersensitivity to any of the excipients contained in the study drug formulation.
* Any other criteria (such as a clinically significant screening blood test result), which in the opinion of the Investigator causes the participant not to qualify for the study.
* Evidence of cerebrovascular dementia with a Hachinski score of 4 or more.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
ADAS-Cog (Alzheimer Disease Assessment Scale-Cognition) | 48 weeks
  Reduction in cognitive decline assessed from baseline over 48 weeks with ANAVEX2-73 compared to placebo using the Alzheimer Disease Assessment Scale-Cognition (ADAS-Cog)
ADCS-ADL (Activities of Daily Living) | 48 weeks
  Reduction in decline of the ability to perform daily activities assessed from baseline over 48 weeks with ANAVEX2-73 compared to placebo using the Activities of Daily Living Scale (ADCS-ADL)

SECONDARY OUTCOMES:
CDR-SB (Clinical Dementia Rating Scale Sum of Boxes) | 48 weeks
  Reduction in cognitive decline assessed from baseline over 48 weeks with ANAVEX2-73 compared with placebo using the Clinical Dementia Rating Scale Sum of Boxes (CDR-SB)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 48 weeks
  Assess the safety and tolerability of ANAVEX2-73 compared to placebo

OTHER OUTCOMES:
Number of participants with change of brain volume assessed by MRI | 48 weeks
  To evaluate the effect of ANAVEX2-73 on structural and Arterial Spin Labeling (ASL) MRI scan assessments characteristic for AD pathophysiology compared to placebo over a 48-week treatment duration
Blood assessment | 48 weeks
  Blood assessment from baseline and compared to placebo at +48 weeks: Abeta40, Abeta42, T-tau, NFL, YKL-40, BACE1 concentration
CSF assessment | 48 weeks
  Changes in CSF parameters (Abeta40, Abeta42, T-tau, P-tau, NFL, YKL-40, neurogranin, BACE1 concentration) characteristic for AD pathophysiology from baseline and compared to placebo at
  +48 weekstreatment differences within subgroups will be performed
Number of participants with pre-specified genetic variants | 48 weeks
  AD relevant pre-specified genetic variants will be assessed. Statistical testing of treatment differences within subgroups will be performed
RSCAQ sleep score | Weeks 0, 4, 12, 24, 36, and 48
  To evaluate whether ANAVEX2-73 improves sleep continuity as assessed on a serial basis (weeks 0, 4, 12, 24, 36, and 48) with a questionnaire that assess reported sleep continuity (RSCAQ)

CONTACTS AND LOCATIONS:
Locations (54):
- Australia (16):
  - Central Coast Neurosciences Research, Central Coast, New South Wales
  - Hornsby (Northern Sydney Health), Hornsby, New South Wales
  - KaRa MINDS, Macquarie Park, New South Wales
  - St Vincent Hospital Sydney, Sydney, New South Wales
  - University of Sydney, Sydney, New South Wales
  - Gold Coast Memory Disorders Clinic, Southport, Quennsland
  - The Royal Adelaide Hospital (RAH) and The Queen Elizabeth Hospital (TQEH), Adelaide, South Australia
  - Penninsula Therapeutic and Research Group, Frankston, Victoria
  - Geelong Private Medical Centre, Geelong, Victoria
  - Delmont Private Hospital, Glen Iris, Victoria
  - Hammond Care, Malvern, Victoria
  - Alfred Health, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Monash Alfred Psychiatry Research Centre, Melbourne, Victoria
  - Royal Melbourne Hospital (RMH), Parkville, Victoria
  - McCusker, Nedlands, Western Australia
- Canada (11):
  - Healthy Brain Aging Labs Uni of Calgary, Calgary, Alberta
  - University of British Columbia Hospital, Vancouver, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - True North Clinical Research, Halifax, Nova Scotia
  - True North Clinical Research, Kentville, Nova Scotia
  - Parkwood Institute, London, Ontario
  - Bruyere Continuing Care, Ottawa, Ontario
  - Kawartha Centre, Peterborough, Ontario
  - Bay Crest Health Sciences, Toronto, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
- Germany (8):
  - University of Ulm, Memory Clinic, Ulm, Baden-Wurttemberg
  - Bayreuth Clinic, Hohe Warte Hospital, Bayreuth, Bavaria
  - Technical University of Munich, School of Medicine, München, Bavaria
  - Central Institute of Mental Health, Mannheim, Hesse
  - Goettingen University Medicine, Clinic for Psychiatry and Psychotherapy, Göttingen, Lower Saxony
  - University Hospital, Bonn, Bonn, North Rhine-Westphalia
  - Clinic for Psychiatry and Psychotherapy, Mainz, Rhineland-Palatinate
  - Charite University Medicine, Berlin
- Netherlands (3):
  - Brain Research Center, 's-Hertogenbosch
  - Brain Research Center, Amsterdam
  - Brain Research Center, Zwolle
- United Kingdom (16):
  - MAC Clinical Research, Teesside, County Teesside
  - University of Edinburgh, Edinburgh, Scotland
  - Glasgow Memory Clinic, Glasgow, Scotland
  - Cognition Health, Guildford, Surrey
  - MAC Clinical Research, Barnsley
  - Cognition Health, Birmingham
  - MAC Clinical Research, Blackpool
  - MAC Clinical Research, Cannock
  - MAC Clinical Research, Leeds
  - MAC Clinical Research, Liverpool
  - Cognition Health, London
  - Imperial College, London
  - King's College, London
  - MAC Clinical Research, Manchester
  - Cognition Health, Plymouth
  - Southern Health NHS Foundation Trust, Southampton